CLINICAL TRIAL: NCT06462911
Title: HOme-Based Self-management and COgnitive Training CHanges Lives (HOBSCOTCH) - SPANISH/ESPAÑOL
Brief Title: Epilepsy Self-Management for Spanish Speakers: HOBSCOTCH - ESPANOL
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: The project has been revised and will be considered not human research.
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Responsible Party: Principal Investigator, Elaine T. Kiriakopoulos, Elaine T. Kiriakopoulos, MD, MPH, MSc Assistant Professor of Neurology, Geisel School of Medicine at Dartmouth Director, HOBSCOTCH Institute for Cognitive Health & Well-Being Dartmouth Hitchcock Epilepsy Center, Dartmouth-Hitchcock Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: STUDY02002468
Record Dates: First submitted 2024-05-14; First posted 2024-06-17 (Actual); Last update posted 2024-08-30 (Actual); Status verified 2024-08

CONDITIONS: Epilepsy; Cognitive Dysfunction; Memory Disorders
Keywords: Epilepsy; Memory; Cognitive training; Self management
MeSH Terms: conditions — Epilepsy; Cognitive Dysfunction; Memory Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Spanish speaking participant with self-reported epilepsy and cognitive and memory dysfunction (Experimental): Participants will receive the HOBSCOTCH intervention (in Spanish) consisting of 1:1 sessions delivered once per week including:
  1 pre-HOBSCOTCH Session (on webcam or by phone)
  1 educational session (on webcam) 6 HOBSCOTCH intervention sessions (webcam or phone)
  1 wrap-up session (webcam or phone)
  Interventions: Behavioral: HOme-Based Self-management and COgnitive Training CHanges lives (HOBSCOTCH) - Spanish/Espanol

INTERVENTIONS:
Behavioral: HOme-Based Self-management and COgnitive Training CHanges lives (HOBSCOTCH) - Spanish/Espanol — HOBSCOTCH is a home-based self-management program to treat cognitive symptoms and improve quality of life, while minimizing the barriers of access to care. The program is based on Problem Solving Therapy (PST) and teaches problem solving strategies and compensatory mechanisms to help manage cognitive dysfunction and enhance quality of life. The entire HOBSCOTCH program has been translated into Spanish for people with epilepsy who speak Spanish.
  Other Names: HOBSCOTCH-Spanish/Espanol

SUMMARY:
The goal of this pilot study is to assess the feasibility of translating and delivering the existing home-based epilepsy self-management intervention, HOBSCOTCH, for people with epilepsy whose primary language is Spanish.

The main questions it aims to answer are:

1. Can the current HOBSCOTCH program be successfully translated for Spanish speaking people with epilepsy?
2. Will people with epilepsy who speak Spanish experience improved quality of life similar to that found in people with epilepsy who received the HOBSCOTCH program in English?

Participants will be asked to:

* attend nine, one-hour virtual (online and/or by telephone) HOBSCOTCH-SPANISH sessions with a one-on-one certified bilingual HOBSCOTCH coach
* complete a brief clinical questionnaire about their diagnosis of epilepsy
* complete two questionnaires before and after the HOBSCOTCH sessions about their quality of life and about memory and thinking processes
* keep a short daily diary about their seizures, symptoms and use of the self-management strategies taught in the HOBSCOTCH program
* complete a brief Satisfaction Survey and a 3 question survey about shared decision making after the entire HOBSCOTCH program

ELIGIBILITY:
Inclusion Criteria:

* Adult (18 + years)
* Self-reported epilepsy with controlled or uncontrolled seizures
* Spanish as primary language
* Literate in Spanish (per bilingual Cognitive Coach)
* Access to the internet and/or a telephone

Exclusion Criteria:

* Self-report of a dementing illness, a dementing illness appearing in their medical record if available or in the judgment of the Principal Investigator or Bilingual Coach
* Severe mental disability or estimated IQ less than 70 per clinical judgement of the Principal Investigator or Bilingual Coach
* Significant visual impairment precluding reading or writing
* No reliable telephone or internet access
* No self-reported diagnosis of epilepsy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-09 (Estimated); Primary Completion 2025-01 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
Change in quality of life as measured by comparing the pre and post HOBSCOTCH-Spanish/Espanol intervention scores on the Quality of Life in Epilepsy-10 (QOLIE-10). | Before the HOBSCOTCH program and after the HOBSCOTCH program, approximately 9 weeks later.
  The QOLIE-10 is a standard, brief questionnaire that asks people with epilepsy about the impact of their condition on their lives. It consists of 10 questions based on a 5-point Likert scale ranging from "none of the time or not at all" to "all of the time or extremely." The scoring ensures that positive responses are represented by lower numbers, while negative responses correspond to higher numbers. The total score is calculated by summing the scores for all answered questions and dividing by the number of items answered. Patients with lower scores experience fewer problems related to their epilepsy.
Change in subjective cognition as measured by comparing the pre and post HOBSCOTCH-Spanish/Espanol intervention scores on NeuroQOL - Cognitive Function sub-scale. | Before the HOBSCOTCH program and after the HOBSCOTCH program, approximately 9 weeks later.
  The Cognitive Function sub-scale of the NeuroQOL is a brief validated tool developed by the NIH for use in patients with neurological disease. Scores range from 8 to 40, with a higher score indicating better reported cognitive functioning.

SECONDARY OUTCOMES:
Participant satisfaction with the HOBSCOTCH-Spanish/Espanol program as measured by analyzing a Participant Satisfaction Survey at the end of the study. | After the completion of the HOBSCOTCH-Spanish/Espanol program, approximately 9 weeks later.
  The Participant Satisfaction Survey has been developed through the original HOBSCOTH program and is used in clinical practice for quality improvement and was translated into Spanish. It contains 10 items scored on a 5-point Likert scale with a higher score indicating greater satisfaction with the program.
Evaluation of participants' perception of shared-decision making during HOBSCOTCH-Spanish/Espanol intervention as measured by CollaboRATE score. | After the completion of the HOBSCOTCH-Spanish/Espanol program, approximately 9 weeks later.
  CollaboRATE is a brief patient survey focused on shared decision making. It employs a 3-item assessment of patient perception of how much effort was made to hear, understand and incorporate their concerns into the program. The items are measured on a 10-point Likert scale in which 0 indicates that no effort was made and 9 indicates every effort was made. Higher scores indicate a greater degree or positive impression of patient perception of shared decision making.

CONTACTS AND LOCATIONS:
Overall Officials: Elaine T Kiriakopoulos, MD, MPH, MSc, Principal Investigator — Dartmouth-Health/Dartmouth-Hitchcock, Dartmouth College
Locations (1):
- Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire, United States